CLINICAL TRIAL: NCT01123538
Title: Progestagen Type in Postmenopausal Hormone Therapy and Blood Gene Expression
Brief Title: Progestagen Type in Postmenopausal Hormone Therapy and Blood Gene Expression Profile
Acronym: ProGEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EudraCT-2006-004462-14; 2006-004462-14 (EudraCT Number)
Record Dates: First submitted 2010-04-30; First posted 2010-05-14 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacogenomics; Systems Biology
MeSH Terms: interventions — Progesterone; Chlormadinone Acetate

ARMS (2):
- Natural progesterone (Other): Combined menopausal treatment containing natural progesterone
  Interventions: Drug: Progesterone
- Chlormadinone acetate (Active Comparator): Combined menopausal treatment containing chlormadinone acetate
  Interventions: Drug: Chlormadinone acetate

INTERVENTIONS:
Drug: Progesterone — 200 mg/day oral micronized natural progesterone (e.g. Utrogestan® 100mg) + 0.05 mg/day transdermal (i.e. plaster) 17β-estradiol (e.g. Estraderm® 50µg) during a year
  Arms: Natural progesterone
Drug: Chlormadinone acetate — 5 mg/day oral chlormadinone acetate (e.g. Luteran® 5mg)+ 0.05 mg/day transdermal (i.e. plaster) 17β-estradiol (e.g. Estraderm® 50µg)
  Arms: Chlormadinone acetate

SUMMARY:
The purpose of this study is to compare combined postmenopausal hormone therapy natural progesterone to the one containing synthetic progestagen (i.e. chlormadinone acetate) at the blood transcriptome level.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women defined as:

  * 45 years< age < 65 years
  * Amenorrhoeic for ≥ 1 year
  * Amenorrhoeic for < 1 year either without any withdrawal vaginal bleeding for 3 consecutive months in spite of a cyclic progestagen treatment and/or blood estradiol levels ≤ 20 pg/mL and blood FSH levels ≥ 40 UI/mL
  * Women with bilateral ovariectomy
* Women suffering of at least 1 postmenopausal symptoms listed:

  * Hot flashes,
  * Memory and Concentration Problems,
  * Mood Swings,
  * Insomnia,
  * Urinary Incontinence,
  * Night sweating,
  * Join pains,
  * Asthenia.
* No use of hormone therapy (HT)
* Previous HT user:

  * HT use < 3 months - stop for 6 months
  * HT use <= 1 year - stop for > 12 months
* If previous use of soya derivatives in dietary supplements: washout period = 3 months
* Signed informed consent, after having received both oral- and written- information regarding the study goals, its risks and benefits and its constraints, including the 12 month follow-up. A delay should be respected between information and the signature of the written consent.

Exclusion Criteria:

* Past HT users who have used treatment for more than 1 year
* Hysterectomized women
* Women without health insurance (only in French centre)
* History of cardio-vascular accident either arterial or venous
* Untreated high blood pressure
* Liver disease
* Diabetes
* History of cancer except basal-cell skin cancer and colon cancer
* Severe history of familial breast cancer defined as at least 2 women first degree- relatives with breast cancer diagnosis before 50 years
* History of severe mastalgia
* History of breast biopsy showing hyperplasia (with or without atypia)
* Undiagnosed vaginal bleeding
* Diagnosed endometrial hyperplasia
* Auto-immune disease (e.g. lupus)
* Women with kidney transplant

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Whole blood and white blood cells gene expression profiling after 3 months of HT treatment | 0 and 3 months after treatment

SECONDARY OUTCOMES:
Quality of life, proteome, plasma haemostatic variable measurements | 0,3,6 and 12 months
Whole blood and white blood cells gene expression profiling after 12 months of HT treatment | 0 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eiliv Lund, MD, PhD, Principal Investigator — Institute of Community Medicine, Tromsø, Norway; Vanessa Dumeaux, PharmD, PhD, Study Director — Institute of community medicine, Tromsø, Norway
Locations (1):
- Gynecology center, Helse Nord, Bodø, Norway